CLINICAL TRIAL: NCT05084508
Title: A Phase II, Observer-blind, Randomized, Controlled Study to Evaluate the Immunogenicity and Safety of a Varicella Vaccine at Various Potencies Compared With Varivax, as a First Dose, Administered in Healthy Children in Their Second Year of Life
Brief Title: A Study on the Immune Response and Safety of Various Potencies of an Investigational Chickenpox Vaccine Compared With a Marketed Chickenpox Vaccine, Given to Healthy Children 12 to 15 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 217212; 2022-001910-21 (EudraCT Number)
Record Dates: First submitted 2021-10-18; First posted 2021-10-19 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Chickenpox
Keywords: Varicella; Chickenpox
MeSH Terms: conditions — Chickenpox | interventions — Measles-Mumps-Rubella Vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Observer-blind study. Recipients and study evaluators will be unaware of vaccine administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- VNS_Low Group (Experimental): Participants received 1 dose of an investigational varicella vaccine (VNS) of low potency, 1 dose of a measles, mumps, and rubella (MMR) vaccine, 1 dose of a hepatitis A vaccine (Havrix) and 1 dose of a13 valent pneumococcal conjugate vaccine (Prevnar 13) on Day 1.
  Interventions: Biological: Investigational varicella vaccine low potency; Biological: Measles, mumps, and rubella vaccine; Biological: Hepatitis A vaccine; Biological: 13-valent pneumococcal conjugate vaccine
- VNS_Med Group (Experimental): Participants received 1 dose of VNS vaccine of medium potency, 1 dose of MMR vaccine, 1 dose of Havrix vaccine, and 1 dose of Prevnar 13 vaccine on Day 1.
  Interventions: Biological: Investigational varicella vaccine medium potency; Biological: Measles, mumps, and rubella vaccine; Biological: Hepatitis A vaccine; Biological: 13-valent pneumococcal conjugate vaccine
- VNS_High Group (Experimental): Participants received 1 dose of VNS vaccine of high potency, 1 dose of MMR vaccine, 1 dose of Havrix vaccine, and 1 dose of Prevnar 13 vaccine on Day 1.
  Interventions: Biological: Investigational varicella vaccine high potency; Biological: Measles, mumps, and rubella vaccine; Biological: Hepatitis A vaccine; Biological: 13-valent pneumococcal conjugate vaccine
- VV_Lot1 and Lot2 Pooled Group (Active Comparator): Participants received 1 dose of a licensed varicella vaccine (VV) of Lot 1 or 1 dose of a licensed vaccine (VV) of Lot 2, 1 dose of MMR vaccine, 1 dose of Havrix vaccine, and 1 dose of Prevnar 13 vaccine on Day 1.
  Interventions: Biological: Licensed varicella vaccine Lot 1; Biological: Licensed varicella vaccine Lot 2; Biological: Measles, mumps, and rubella vaccine; Biological: Hepatitis A vaccine; Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: Investigational varicella vaccine low potency — 1 dose of a low-potency investigational varicella vaccine administered subcutaneously.
  Arms: VNS_Low Group
Biological: Investigational varicella vaccine medium potency — 1 dose of a medium-potency investigational varicella vaccine administered subcutaneously.
  Arms: VNS_Med Group
Biological: Investigational varicella vaccine high potency — 1 dose of a high-potency investigational varicella vaccine administered subcutaneously.
  Arms: VNS_High Group
Biological: Licensed varicella vaccine Lot 1 — 1 dose of a licensed varicella vaccine of Lot 1 administered subcutaneously.
  Arms: VV_Lot1 and Lot2 Pooled Group
Biological: Licensed varicella vaccine Lot 2 — 1 dose of a licensed varicella vaccine of Lot 2 administered subcutaneously.
  Arms: VV_Lot1 and Lot2 Pooled Group
Biological: Measles, mumps, and rubella vaccine — 1 dose of a measles, mumps, and rubella vaccine administered subcutaneously.
Biological: Hepatitis A vaccine — 1 dose of a hepatitis A vaccine administered intramuscularly.
Biological: 13-valent pneumococcal conjugate vaccine — 1 dose of a 13-valent pneumococcal conjugate vaccine administered intramuscularly.

SUMMARY:
The purpose of this study is to assess immune response and safety of various potencies of an investigational chickenpox vaccine given to healthy children 12 to 15 months of age.

DETAILED DESCRIPTION:
The study aims to demonstrate the immunogenicity of the investigational VNS vaccine at three potencies (VNS_Low, VNS_Med, and VNS_High) compared to the licensed varicella vaccine, Varivax (VV), as a first dose for children aged 12 to 15 months in the US. To ensure more representative data, participants in the VV group are randomized into two lots (VV_Lot1 and VV_Lot2), which are analyzed as pooled lots throughout the study. Besides assessing immunogenicity, the study also seeks to generate safety data.

In the US, participants will receive additional vaccines: a measles, mumps, and rubella vaccine (MMR), a hepatitis A vaccine (Havrix), and a 13-valent pneumococcal conjugate vaccine (Prevnar 13). Participants outside the US will receive an MMR vaccine (M-M-R II or M-M-RVaxPro, depending on the country), Havrix, and, in some cases, Prevnar 13, but only in countries where it's recommended for children 12-15 months according to local immunization schedules.

At the end of the study, or shortly after, GSK provided re-vaccination with a dose of Varivax (VV) to participants who did not meet the pre-specified seroresponse threshold of anti-gE antibody concentration was greater than or equal to (>=) 300 mIU/mL. Additionally, a second dose of VV and/or Havrix was offered to participants in non-US countries where local health departments do not routinely provide varicella and/or hepatitis A vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female between, and including, 12 and 15 months of age (i.e., from his/her 1 year birthday until the day before age of 16 months) at the time of the administration of the study interventions.
* Written informed consent obtained from the parent(s)/legally authorized representative(s) of the participant prior to performance of any study-specific procedure.
* Participants' parent(s)/legally authorized representative(s), who, in the opinion of the investigator, can and will comply, with the requirements of the protocol (e.g., completion of Electronic Diaries, return for follow-up visits).
* Only for US participants and participants in countries where pneumococcal conjugate vaccine is recommended at 12-15 months of life as per national immunization schedule: Participants who previously received the primary series of pneumococcal conjugate vaccine in their first year of life with the last dose at least 60 days prior to study entry.

Exclusion Criteria:

Medical Conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions including hypersensitivity to neomycin or gelatin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Hypersensitivity to latex.
* Major congenital defects, as assessed by the investigator.
* History of varicella.
* Recurrent history of or uncontrolled neurological disorders or seizures.
* Participant with history of SARS-CoV-2 infection who is still symptomatic.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior and Concomitant Therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study interventions during the period beginning 30 days before the dose of study interventions (Day -29 to Day 1), or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants, or other immune-modifying drugs during the period starting 90 days prior to the study interventions administration. For corticosteroids, this will mean prednisone equivalent ≥ 0.5 mg/kg/day or 20 mg/day whichever is the maximum dose for pediatric participants, or equivalent. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 180 days before the dose of study interventions or planned administration during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
* Previous vaccination against measles, mumps, rubella, hepatitis A, and/or varicella virus.

Medical Conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions including hypersensitivity to neomycin or gelatin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Hypersensitivity to latex.
* Major congenital defects, as assessed by the investigator.
* History of varicella.
* Recurrent history of or uncontrolled neurological disorders or seizures.
* Participant with history of SARS-CoV-2 infection who is still symptomatic.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior and Concomitant Therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study interventions during the period beginning 30 days before the dose of study interventions (Day -29 to Day 1), or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants, or other immune-modifying drugs during the period starting 90 days prior to the study interventions administration. For corticosteroids, this will mean prednisone equivalent ≥ 0.5 mg/kg/day or 20 mg/day whichever is the maximum dose for pediatric participants, or equivalent. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 180 days before the dose of study interventions or planned administration during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
* Previous vaccination against measles, mumps, rubella, hepatitis A, and/or varicella virus.
* Previous administration of a booster dose of any pneumococcal conjugate vaccine.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the dose and ending at 43 days after the dose of study interventions administration* (Visit 3) with the exception of inactivated influenza (flu) vaccine which may be given at any time during the study and administered at a different location than the study interventions.
* Any other age appropriate vaccine may be given starting at Visit 3 and anytime thereafter.

  * In case of emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor/designee is notified accordingly.

Prior/Concurrent Clinical Study Experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non investigational intervention (drug/invasive medical device).

Other Exclusions

* Child in care.
* Any study personnel's immediate dependents, family, or household members.
* Participants with the following high-risk individuals in their household:

  * Immunocompromised individuals.
  * Pregnant women without documented history of varicella.
  * Newborn infants of mothers without documented history of varicella.
  * Newborn infants born <28 weeks of gestation.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (40):
  - GSK Investigational Site, Bryant, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bellflower, California
  - GSK Investigational Site, Downey, California
  - GSK Investigational Site, Foothill Ranch, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Bridgeton, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Fort Washington, Pennsylvania
  - GSK Investigational Site, Barnwell, South Carolina
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Dickinson, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, Pflugerville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Marshfield, Wisconsin
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Poland (2):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Torun
- GSK Investigational Site, San Juan, Puerto Rico
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- GSK Investigational Site, Ohio, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 800 participants enrolled, 9 participants discontinued before receiving the vaccination and therefore only 791 participants were included in the Exposed Set and started the study.
Pre-assignment Details: * The Prevnar 13 vaccine was administered only to participants enrolled in the US and in countries where pneumococcal conjugate vaccine is recommended at 12- 15 months as per national immunization schedule.
  * As described in the protocol and analysis plan, participants in the varicella vaccine (VV) group are randomized into two lots (VV_Lot1 and VV_Lot2) and analyzed as pooled throughout the study.
Period: Overall Study
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
Started | 203 | 195 | 203 | 190
Completed | 197 | 190 | 193 | 185
Not Completed | 6 | 5 | 10 | 5
Not completed — Lost to Follow-up | 6 | 3 | 7 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 1
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group | Total
Number analyzed (Participants) | 203 | 195 | 203 | 190 | 791
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 203 | 195 | 203 | 190 | 791
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 102 | 101 | 107 | 424
  Male | 89 | 93 | 102 | 83 | 367
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 71 | 74 | 73 | 293
  Not Hispanic nor Latino | 128 | 124 | 128 | 117 | 497
  Missing | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Anti-varicella Zoster Virus (VZV) Glycoprotein E (gE) Antibodies
Description: Concentrations of anti-VZV gE antibodies were presented as Geometric Mean Concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL) for each group.
Time Frame: At Day 43
Population: The analysis was performed on the Per Protocol Set (PPS), which included participants who received all study interventions as per protocol, were not unblinded, had immunogenicity results post-dose, complied with blood draw intervals, without intercurrent medical conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: mlU/ml
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
Number analyzed (Participants) | 171 | 159 | 158 | 161
mlU/ml | 960 [843 to 1093] | 1071 [952 to 1204] | 1555 [1407 to 1718] | 1284 [1136 to 1453]

2. Secondary Outcome: Percentage of Participants With Seroresponse to VZV gE
Description: Seroresponse was defined as the percentage of participants for whom the post-dose of anti VZV gE antibody concentration was greater than or equal to (>=) 300 mIU/mL for each group.
Time Frame: At Day 43
Population: The analysis was performed on the PPS, which included participants who received all study interventions as per protocol, were not unblinded, had immunogenicity results post-dose, complied with blood draw intervals, without intercurrent medical conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
Number analyzed (Participants) | 171 | 159 | 158 | 161
Percentage of participants | 93.6 [88.78 to 96.75] | 96.2 [91.97 to 98.60] | 98.7 [95.50 to 99.85] | 98.1 [94.65 to 99.61]

3. Secondary Outcome: Number of Participants Reporting Each Solicited Administration Site Events
Description: Assessed solicited administration site events included injection site redness, pain and swelling.
Time Frame: Day 1 (post dose) to Day 4
Population: The analysis was performed on the Exposed set (ES), which included all participants who received a study intervention. Analysis per group was based on the varicella intervention administered.
Measure: Count of Participants; unit: Participants
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
Number analyzed (Participants) | 203 | 195 | 203 | 190
Participants
  Injection site pain | 76 | 64 | 70 | 57
  Redness at injection site | 24 | 23 | 35 | 23
  Swelling at injection site | 14 | 11 | 15 | 12

4. Secondary Outcome: Number of Participants Reporting Each Solicited Systemic Events
Description: Solicited systemic events included fever, varicella like rash (including injection site varicella-like rash), and general rash (not varicella-like) after the administration of all vaccines for each group. Fever was defined as temperature >= 38.0 °C (100.4°F) by any route (the preferred location for measuring temperature is the axilla). A typical varicella-like rash manifests as a rash/lesion that may appear within several weeks after the varicella vaccination. Lesions may contain spots, bumps, blisters, or crusts. Includes injection site varicella-like rash.
Time Frame: Day 1 (post dose) to Day 43
Population: The analysis was performed on the ES, which included all participants who received a study intervention. Analysis per group was based on the varicella intervention administered.
Measure: Count of Participants; unit: Participants
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
Number analyzed (Participants) | 203 | 195 | 203 | 190
Participants
  Fever | 49 | 48 | 59 | 44
  Any varicella-like rash | 33 | 31 | 35 | 29
  Any general rash | 66 | 51 | 68 | 59

5. Secondary Outcome: Number of Participants Reporting Each Solicited Systemic Events
Description: Solicited systemic events included drowsiness, loss of appetite, and irritability after the administration of all vaccines for each group.
Time Frame: Day 1 (post dose) to Day 15
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
Number analyzed (Participants) | 203 | 195 | 203 | 190
Participants
  Any drowsiness | 86 | 68 | 93 | 80
  Any loss of appetite | 69 | 57 | 71 | 60
  Any irritability | 112 | 94 | 112 | 109

6. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events
Description: Unsolicited adverse events (AEs) included any AE reported in addition to solicited events during the study, or any "solicited" symptoms with onset outside of the specified period of follow-up for solicited symptoms; these were assessed for each group after the administration of all vaccines. Unsolicited AEs included both serious and non-serious AEs.
Time Frame: Day 1 (post dose) to Day 43
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
Number analyzed (Participants) | 203 | 195 | 203 | 190
Participants | 67 | 53 | 64 | 61

7. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: A SAE was defined as an AE which was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, or other situations that were considered serious per medical or scientific judgment.
Time Frame: From Day 1 to Day 181 (Study end)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
Number analyzed (Participants) | 203 | 195 | 203 | 190
Participants | 2 | 4 | 4 | 6

ADVERSE EVENTS:
Time Frame: SAEs were collected from Day 1 to Day 181 (Study end), solicited administration site events from Day 1 to Day 4, solicited systemic events (drowsiness, loss of appetite and irritability) from Day 1 to Day 15, solicited systemic events and unsolicited AEs (fever, varicella-like rash [including injection site varicella like rash] and general rash [not varicella-like]) from Day 1 to Day 43
Arm/Group | VNS_Low Group | VNS_Med Group | VNS_High Group | VV_Lot1 and Lot2 Pooled Group
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/195 | 0/203 | 0/190
Serious Adverse Events (participants affected / at risk) | 2/203 | 4/195 | 4/203 | 6/190
Other Adverse Events (participants affected / at risk) | 173/203 | 165/195 | 178/203 | 158/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS_Low Group (N=203) | VNS_Med Group (N=195) | VNS_High Group (N=203) | VV_Lot1 and Lot2 Pooled Group (N=190)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS_Low Group (N=203) | VNS_Med Group (N=195) | VNS_High Group (N=203) | VV_Lot1 and Lot2 Pooled Group (N=190)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 4 (4) | 2 (2) | 5 (5)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 7 (7) | 1 (1) | 8 (9) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 5 (8)
Administration site erythema (General disorders) | 24 (40) | 23 (33) | 35 (44) | 23 (31)
Administration site pain (General disorders) | 76 (103) | 65 (82) | 70 (87) | 57 (67)
Administration site swelling (General disorders) | 14 (21) | 11 (16) | 15 (18) | 12 (14)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 49 (99) | 48 (91) | 59 (145) | 44 (87)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Candida nappy rash (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laryngotracheitis obstructive (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 9 (11)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 7 (7) | 1 (2) | 2 (2) | 5 (5)
Otitis media acute (Infections and infestations) | 9 (10) | 6 (6) | 2 (2) | 6 (7)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Roseola (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 6 (6) | 13 (14) | 10 (11)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Torus fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 71 (206) | 57 (131) | 71 (192) | 60 (138)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 87 (217) | 68 (170) | 93 (264) | 80 (174)
Irritability (Psychiatric disorders) | 113 (397) | 94 (278) | 112 (417) | 110 (336)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 5 (5) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 1 (1) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (7) | 5 (5) | 6 (7)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Rash scarlatiniform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rashes, eruptions and exanthems NEC (Skin and subcutaneous tissue disorders) | 76 (443) | 64 (329) | 75 (514) | 72 (350)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT05084508/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT05084508/SAP_001.pdf